CLINICAL TRIAL: NCT07140510
Title: Effectiveness of Dinalbuphine Sebacate in Postoperative Pain Control Following Total Knee Arthroplasty: A Randomized Double Blinded Placebo-controlled Trial
Brief Title: Dinalbuphine Sebacate in Postoperative Pain Control After TKA
Acronym: Naldebain
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Thammasat University (Other)
Responsible Party: Principal Investigator, Supakit Kanitnate, Principal investigator, Thammasat University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OrthoTU14
Record Dates: First submitted 2025-08-03; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Osteo Arthritis of the Knee; Total Knee Anthroplasty
Keywords: Dinalbuphine Sebacate; Naldebain; Subacute pain; postoperative pain; total knee arthroplasty
MeSH Terms: conditions — Pain, Postoperative | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dinalbuphine Sebacate (Experimental): Naldebain 150mg/2mL IM
  Interventions: Drug: Dinalbuphine Sebacate
- Placebo (Placebo Comparator): Normal saline 2 mL IM
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Dinalbuphine Sebacate — Dinalbuphine Sebacate 150 mg intramuscular injection after spinal anesthesia and adductor canal block in the same side of TKA
  Arms: Dinalbuphine Sebacate
Drug: Normal Saline — Normal saline 2 mL intramuscular injection after spinal anesthesia and adddutor canal block
  Arms: Placebo

SUMMARY:
To evaluate the effectiveness of Dinalbuphine Sebacate for controlling subacute pain after total knee arthroplasty

DETAILED DESCRIPTION:
A single dose of intramuscular Dinalbuphine Sebacate can mitigate pain for up to 1 week after TKA

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritic knee patients underwent unilateral primary TKA
* Age 50-90 years
* ASA class I-III
* Participants understand and consent to the protocol of the trial

Exclusion Criteria:

* Morbid obesity (BMI>40)
* Knee osteoarthritis from inflammatory knee arthritis, trauma, infection
* Previous knee surgery
* Cognitive disorder
* Liver disease
* Allergy to NSAIDs, opioids, sesame oil, and benzyl benzoate
* CYP3A4 inhibitor and inducer drugs used

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Visual analog scale for pain (VAS 0-100) | Record every 12 hours after surgery until 2 weeks postoperatively, then once weekly until 12 weeks postopertively
  Visual analog scale for pain at rest and on motion (knee flexion 90 degrees) using 0-100 mm, where a score of 0 represented no pain and 100 indicated the most severe pain

SECONDARY OUTCOMES:
The amount of analgesic drug used | During hospitalization and at home until 12 weeks after surgery
  The amount of IV morphine and oral tramadol (milligram)
Adverse effects | The first week after surgery
  Incidence of adverse effects including pyrexia, nausea, vomiting, dizziness, injection site pain, and somnolence
Length of stay | During hospitalization (from admission to discharge)
  Length of stay (day)
Modified WOMAC score | At pre-operative, 2 weeks, 6 weeks, and 12 weeks postoperatively
  Modified Western Ontario and McMaster Universities Osteoarthritis Index score, including total & subscore. Each item was scored with a Likert scale (0-4). The overall MOWAC was 0-96 (high score = worse symptoms)
Forgotten Joint Score | At pre-operative, 2 weeks, 6 weeks, and 12 weeks postoperatively
  Forgotten Joint Score (Thai version) with 12 questions. Each item was scored on a Likert scale (0-4). The raw score was converted to a 0-100 scale (0 = worst, 100 = best)
Time up and go (TUG) test | At pre-operative, 2 weeks, 6 weeks, and 12 weeks postoperatively
  Time up and go (TUG) test records the time in seconds when the patient starts standing up from the chair, then walks 3 meters at a normal pace, and turns around to sit on the chair.
Knee range of motion | At pre-operative, 2 weeks, 6 weeks, and 12 weeks postoperatively
  Angle of knee flexion and extension in degrees using a long goniometer

OTHER OUTCOMES:
Rate of closed manipulation | At 3 months postoperatively
  Closed manipulation under anesthesia due to an unsatisfactory range of motion

CONTACTS AND LOCATIONS:
Locations (1):
- Thammasat University, Khlong Luang, Changwat Pathum Thani, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yeh CY, Jao SW, Chen JS, Fan CW, Chen HH, Hsieh PS, Wu CC, Lee CC, Kuo YH, Hsieh MC, Huang WS, Chung YC, Liou TY, Chiu HH, Tseng WK, Lee KC, Wang JY. Sebacoyl Dinalbuphine Ester Extended-release Injection for Long-acting Analgesia: A Multicenter, Randomized, Double-Blind, And Placebo-controlled Study in Hemorrhoidectomy Patients. Clin J Pain. 2017 May;33(5):429-434. doi: 10.1097/AJP.0000000000000417. PMID 27518486